CLINICAL TRIAL: NCT06179797
Title: Chronic Remote Ischemic Conditioning in Vascular Cognitive Impairment: A Dose Escalation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Collaborators: Georgia Rehabilitation Institute (Unknown)
Responsible Party: Principal Investigator, Askiel Bruno, MD, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1513705-3
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Age-related Cerebral White Matter Changes; Cognition Disorder
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: concealed allocations and blinded laboratory personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- sham (Sham Comparator): BP cuff bilateral arm compression to 50 mmHg.
  Interventions: Device: remote ischemic conditioning
- dose 1 (Active Comparator): BP cuff bilateral arm compression to 50 mmHg above systolic BP for 2.5 minutes on/off for 4 cycles every other day.
  Interventions: Device: remote ischemic conditioning
- dose 2 (Active Comparator): BP cuff bilateral arm compression to 50 mmHg above systolic BP for 5 minutes on/off for 4 cycles every other day.
  Interventions: Device: remote ischemic conditioning
- dose 3 (Active Comparator): BP cuff bilateral arm compression to 50 mmHg above systolic BP for 5 minutes on/off once daily.
  Interventions: Device: remote ischemic conditioning
- dose 4 (Active Comparator): BP cuff bilateral arm compression to 50 mmHg above systolic BP for 5 minutes on/off twice daily.
  Interventions: Device: remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — suprasystolic BP sequential compression of both arms with blood pressure cuffs for 5 min on/off for 4 cycles.
  Other Names: RIC

SUMMARY:
To evaluate the dose-response of relevant blood biomarkers to remote ischemic conditioning in patients with age-related cerebral white matter hyperintensities on MRI, in preparation for a subsequent larger efficacy trial.

DETAILED DESCRIPTION:
Objective: The objective of this early phase study is to evaluate the dose-response of relevant blood biomarkers to remote ischemic conditioning in preparation for a subsequent larger efficacy trial. In addition, we will evaluate the tolerability and adherence to the treatment protocol.

Aim: We aim to measure blood biomarkers in response to daily remote ischemic conditioning (RIC) using a dose escalation study design in 40 patients with age-related cerebral white matter hyperintensities on MRI.

Hypothesis: We hypothesize that there will be a significant change in the biomarker levels in a dose dependent fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥55 years
2. Head MRI in the past 6 months showing no more than moderate age related cerebral white matter changes (Fazekas score 0-2).
3. Able to walk without assistance & independently perform basic activities of daily living.
4. Able to understand this study and agree for a valid consent.

Exclusion Criteria:

Prior non-lacunar (cortical) stroke. 2. Unable to cooperate with the use of the conditioning device. 3. Confounding illness that might interfere with the interpretation of results (such as active malignancy or multiple sclerosis).

4. Contraindication to transient arm ischemia in either arm (such as symptomatic peripheral artery disease).

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
RBC deformability index | 5 weeks total study duration
  from baseline to 4 weeks of treatment and one week off treatment

SECONDARY OUTCOMES:
inflammatory and anti-inflammatory Interleukins | 5 weeks
  ability to tolerate and adhere to protocol treatments.
tolerability | 4 weeks
  any discontinuation and adverse events during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Smith, RN, Study Director — Wellstar MCG Health
Locations (1):
- Wellstar MCG Health, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
yes, upon reasonable request.